CLINICAL TRIAL: NCT05255367
Title: Impact of the Consumption of (Poly)Phenolic Rich Products on Cardiometabolic Risk Markers in Postmenopausal Women
Brief Title: Effect of (Poly)Phenolic on Cardiometabolic Risk of Postmenopausal Women
Acronym: CARDIOGENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Mª Jesús Periago, PhD, Full Professor of Nutrition and Food Science, Universidad de Murcia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: (Poly)phenol and menopause; 20904/PI/2018 (Other Grant/Funding Number: Fundación Séneca (Research Agency of Murcia, Spain))
Record Dates: First submitted 2022-01-10; First posted 2022-02-24 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Post-menopausal Women; Overweight and Obesity
Keywords: Menopause; (Poly)phenols; Cardiometabolic risk; Oxidative stress; Lipid and glucose metabolism
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intake of (poly)phenol rich foods (Experimental): Daily consumption of 100 ml of a commercial juice of berries and pomegranate, 20 g dark chocolate and 1 green tea, to test if the supplementation of the diet with (poly)phenol rich foods, during 2 months, reduce the cardiometabolic risk in post-post-menopausal women.
  Interventions: Combination Product: (poly)phenols rich foods

INTERVENTIONS:
Combination Product: (poly)phenols rich foods — Prior to start the intervention (initial time of the study) the volunteers will follow their habitual diet during 30 days as a control period, and then they will start with the intervention period (baseline) following their habitual diet supplemented with (poly)phenol rich products during 60 days (after intervention).
  At the beginning of the study (initial time), at the beginning of the intervention (baseline) and at the end of the intervention (after the intervention) with rich (poly)phenols foods, biological samples (blood, urine and feces) and anthropometric measurements will be taken. In addition, the participants will record the food intake weekly with a 24 h dietary-recall form.

SUMMARY:
The purpose of this investigation is to test the hypothesis that in post-menopausal women with cardiometabolic risk, eating a relatively high daily amount of (poly)phenol-containing products (green tea, dark chocolate and berries) could reduce the risk of metabolic syndrome and cardiovascular disease. Changes in different biomarkers of lipid metabolism, glucose metabolism, inflammation and oxidative stress will be evaluated. Other related factors may be also affected, such as body mass index (BMI) and the percentage of body fat, dietary habits (total energy intake and macronutrient distribution) and microbiota composition.

DETAILED DESCRIPTION:
Menopause is a stage characterized by the sudden decrease in estrogens linked to the absence of amenorrhea for at least 12 months. Estrogens are involved in certain metabolic pathways such as lipids metabolism and the distribution of body fat in the body. As a result of the fall of estrogen production, postmenopausal women experience a number of alterations of the energy homeostasis that are accompanied by an increase in body weight and a tendency to obesity and visceral fat deposition, as well as variations in the levels of total cholesterol (T-C), low-density lipoprotein-cholesterol (LDL-C), high-density lipoprotein-cholesterol (HDL-C) and triglycerides (TGs), increasing the risk for cardiometabolic diseases. In addition, menopause contributes to disorders of the glucose metabolism increasing insulin resistance (IR) that can predispose to the development of type 2 diabetes mellitus (T2DM).

(Poly)phenols are recognized as bioactive compounds with general antioxidant and anti-inflammatory activity and as potent vasodilators and stimulators of the immune response with the capacity to modulate a range of cardiovascular and metabolic risk factors. An increasing number of intervention studies have built up the evidence of the cardiovascular and metabolic benefits of the intake of these compounds in humans, however, the results remain limited and contradictory, leading to the current controversy regarding the consistency and magnitude of the protective effects that these compounds exert in humans. The lack of consistent and significant results may be partially due to the heterogeneity of the studies and the interindividual variability of the participants.

The investigators have designed this intervention to clearly described the effects of the (poly)phenolic compounds in postmenopausal women with a well-characterized cardiometabolic status. The observed beneficial effects will be correlated with the absorption and metabolism of these compounds.

The protocol will be a single arm intervention study with 22 postmenopausal women as a participants. Prior to start the intervention (initial time of the study) the volunteers will follow their habitual diet during 30 days as a control period. Immediately, they will start with the intervention period (baseline) following their habitual diet supplemented with (poly)phenol rich products, eating daily 100 ml of a commercial juice of berries and pomegranate, 20 g dark chocolate and 1 green tea, during 60 days (after intervention).

At the beginning of the study (initial time), at the beginning of the intervention (baseline) and at the end of the intervention (after the intervention) with rich (poly)phenols foods, biological samples (blood, urine and feces) and anthropometric measurements will be taken. In addition, the participants will record the food intake weekly with a 24 h dietary-recall form.

The investigators will evaluate followed parameters: 1) glucose metabolism indicators, i.e. glucose, insulin and Homeostatic Model Assessment of IR (HOMA-IR), 2) lipid profile (T-C, LDL-C, HDL-C and TGs), 3) blood pressure, both, systolic blood pressure (SBP), and diastolic blood pressure (DBP), 4) biomarkers of inflammation, CRP, TNF-α, adiponectin, soluble vascular cell adhesion molecule 1 (sVCAM-1), soluble intercellular adhesion molecule 1 (sICAM-1), 5) biomarkers of oxidative stress: oxidized isoprostanes and malonaldehyde (MDA), 6) body mass index, body fat and waist-to-hip ratio, 7) dietary habits (total energy intake and macronutrient distribution), 8) metabolites and catabolites of (poly)phenols, and 9) changes in the microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Women 45-65 years old
* With 12 months of amenorrhea
* With overweight or obesity (BMI 25-32) or high percentage of body fat or waist to hip ratio >0.85.
* Total cholesterol lower than 240 mg/dL

Exclusion Criteria:

* Pre-menopausal women
* Hormonal therapy and other pharmacological treatment
* Less than 12 months of amenorrhea
* Smoking women
* Endocrine (Diabetes mellitus or others), renal, hepatic, cancer or psychiatric disorders

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We need women for the study because the aim is to determine the effect of phenolic compounds in postmenopausal women
Enrollment: 26 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in serum levels of glucose and insulin. | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  The investigators will measure the changes in levels of glucose and insulin. samples
Changes in plasmatic lipid profile. | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  the investigators will measure the changes in levels of total cholesterol, LDL-cholesterol, HDL-cholesterol and total triglycerides.
Changes in blood pressure. | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  Both, systolic blood pressure (SBP), and diastolic blood pressure (DBP) will be measure.
Changes in biomarkers of inflammation in plasma. | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  The investigators will measure the CRP, the TNF-α, the adiponectin, the soluble vascular cell adhesion molecule 1 (sVCAM-1) and the soluble intercellular adhesion molecule 1 (sICAM-1).
Changes in biomarkers of oxidative stress in urine. | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  The investigators will measure the level of isoprostanes and malonaldehyde. (MDA)

SECONDARY OUTCOMES:
Changes in body mass index. | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  The investigators will measure the body mass index (Kg/m^2).
Changes in body composition. | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  The investigators will measure the percentage of the body fat mass, body lean mass, total body water and body bone mass using a Tanita DC-430-MA analyzer.
Changes hip-to-waist ratio. | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  The investigators will measure the hip-to-waist ratio.
Dietary habits (total energy intake and macronutrient distribution). | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  The diet will be registered during interventions periods. Volunteers registered the intake of food during 24 h (2 days/week) to determine the adherence to the Mediterranean diet and quantify the intake of energy and macronutrients distribution.

OTHER OUTCOMES:
Changes in the microbiota in feces | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  The investigators will analyze the changes in the diversity and abundance of microbiota to evaluate the prebiotic effect of polyphenols and to understand the bioavailability
Analysis of metabolites and catabolites of (poly)phenols in different biological samples | At initial time of the study, at baseline (the beginning of the intervention) and after 60 days of intake rich (poly)phenols foods (after the intervention)
  The investigators will analyze in urine and feces the metabolites and catabolites of (poly)phenols to evaluate their bioavailability

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Periago Castón, Full Prof., Study Director — Universidad de Murcia; Rocio González Barrio, Assis. Prof., Principal Investigator — Universidad de Murcia
Locations (1):
- Edificio Pleyades-Vitalys 5ª y 6ª planta, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No